CLINICAL TRIAL: NCT00531739
Title: Phase 4 Evaluation of SurgiWrapTM to Minimize Soft Tissue Attachment & Reduce the Incidence of Early Post-Operative Bowel Obstruction in Colorectal Surgery
Brief Title: SurgiWrapTM to Reduce Soft Tissue Attachment & Incidence Early Post-Operative Bowel Obstruction in Colorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cytori Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SURGIWRAP(TM)
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Adhesions; Colectomy
Keywords: Surgery; Colectomy; Proctocolectomy; Adhesions
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (No Intervention): Colorectal Surgery without use of SurgiWrapTM
- B (Active Comparator): Colorectal Surgery with use of SurgiWrapTM film secured in two study areas: the posterior pelvic rim and directly below the abdominal incision
  Interventions: Other: Polylactic Acid Sheet

INTERVENTIONS:
Other: Polylactic Acid Sheet — SurgiWrapTM film will be secured in two study areas: directly below the abdominal incision and on the posterior pelvic rim. The film will not be wrapped directly around an anastomosis.
  Other Names: SurgiWrapTM
  Arms: B

SUMMARY:
The purpose of this study is to determine if the use of SurgiWrapTM: (1) prevents/lowers the incidence of Grade 2 or higher soft tissue attachments under the incision made during abdominal surgery, (2) reduces post-operative bowel obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older of either gender
* Patient has primary diagnosis requiring a two-stage colectomy or procto-colectomy
* Patient or his/her legal representative has read and signed the Institutional Review Board (IRB) approved Informed Consent form before randomization.
* Patient must be able and willing to follow study procedures and instructions.

Exclusion Criteria:

* Patient is participating in another clinical study which may influence adhesion formation.
* Patient has had barriers, solutions, or anti-adhesive therapy, other than SurgiWrapTM, as planned at randomization, placed in the abdomen at the time of the initial surgery
* Patient who, at the initial surgery, had administration of irrigants containing corticosteroids, heparin, salicylates, nonsteroidal anti-inflammatory drugs, or dextran 70
* Patient has one or more medical condition(s), including severe renal, hepatic, hematologic, neurologic, or immune disease that, in the opinion of the Investigator, would make the patient an inappropriate candidate for this study.
* Patient is taking chronic (i.e., > 2 weeks) therapeutic doses of medications known to affect healing such as nonsteroidal anti-inflammatory drugs. Prophylactic aspirin (less than or equal to 325 mg once daily) for cardiovascular indications will be permitted in patients.
* Patient has an infection in the intra-abdominal or pelvic area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-03; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of SurgiWrapTM in the prevention/reduction of Grade 2 or higher soft tissue attachments under the abdominal incision made during colorectal surgery | 6 months

SECONDARY OUTCOMES:
Clinical and radiographic evidence of bowel obstruction | 5 to 30 days
The incidence and extent of soft tissue attachments under the abdominal incision and on the pelvic floor after colorectal surgery | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M Milstein, MD, Study Director — Cytori Therapeutics; Robert Beard, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California Norris Cancer Hospital, Los Angeles, California, United States